CLINICAL TRIAL: NCT05248022
Title: Efficacy and Safety of DEB-BACE Combined With PD-1 Inhibitors in Stage II/III NSCLC With Standard Treatment Failure: A Prospective, Multicenter, Randomized, Open, Double-arm Clinical Trial
Brief Title: Efficacy and Safety of DEB-BACE Combined With PD-1 Inhibitors in Stage II/III NSCLC With Standard Treatment Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Jiangxi Chest Hospital (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJLS-KLDMIR-21002
Record Dates: First submitted 2021-12-17; First posted 2022-02-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung cancer; Drug-eluting Beads Bronchial Arterial Chemoembolization; PD-1 inhibitor; advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is an open-label study. The Participants and investigators are not blinded, but the outcomes assessor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Treatment Group (Experimental): Drug-eluting Beads Bronchial Arterial Chemoembolization combined with Programmed Cell Death Protein 1 Inhibitor was used for treatment.
  Interventions: Procedure: Drug-eluting beads bronchial arterial chemoembolization; Drug: Programmed Cell Death Protein 1 Inhibitor
- Single Treatment Group (Active Comparator): Only receive drug-eluting beads bronchial arterial chemoembolization treatment.
  Interventions: Procedure: Drug-eluting beads bronchial arterial chemoembolization

INTERVENTIONS:
Procedure: Drug-eluting beads bronchial arterial chemoembolization — Drug-eluting beads bronchial arterial chemoembolization generally uses platinum-containing two-drug chemotherapy "platinum (cisplatin, carboplatin, nedaplatin) combined treatment, and drug-loaded microspheres can be loaded with vinorelbine, gemcitabine, irinote Kang, raltitrexed. The dose of chemotherapy drugs is set to 75mg/m2 of platinum, and the dose of chemotherapy through catheter infusion is reduced by 25%. The dose of drug-loaded drugs is vinorelbine 25mg/m2, gemcitabine generally 1000mg/m2, irinotecan 80mg/ m2, raltitrexed 4mg. Chemotherapy was perfused first, followed by embolization with drug-loaded microspheres, until the blood flow in the artery supplying the tumor slowed down and approached stagnation. The number of DEB-BACE treatments is determined by the investigator, and is given as needed according to the patient's condition, usually 1-2 times, with an interval of 28±10 days.
Drug: Programmed Cell Death Protein 1 Inhibitor — Programmed cell death protein 1 inhibitor fixation was treated with sintilimab (Xinda Biopharmaceutical Co., Ltd.). It is administered by intravenous infusion, and the recommended dose is 200 mg, given once every 21 days. The medication will last for two years until disease progression or intolerable toxicity occurs. During immunotherapy, immunosuppressive agents will not be replaced and the dose will not be adjusted.
  Arms: Combination Treatment Group

SUMMARY:
This study is a prospective, multi-center, randomized, open-ended, double-arm clinical study. All eligible patients were randomly assigned to DEB-BACE combined with PD-1 inhibitor (Sindilizumab) treatment group (test group) and DEB-BACE treatment group (control group), to explore the efficacy and safety of combination therapy for stage II/III NSCLC with standard treatment failure or intolerable patients.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old, no gender limit.
* According to the Diagnosis and Treatment of Primary Lung Cancer (2018 edition), non-small cell lung cancer (NSCLC) was diagnosed by histopathology.
* Tumor Node Metastasis (TNM) staging is II-III.
* According to the National Comprehensive Cancer Network (NCCN) guidelines, patients who had failed, refused, or were not suitable for standard treatment (surgery, chemoradiotherapy, targeted) after consultation.
* Eastern Cooperative Oncology Group (ECOG), Performance Status (PS) Score ≤ 2.
* Estimated survival time is more than 3 months.
* The patient has signed informed consent.

Exclusion Criteria:

* The patient has previously received interventional therapy [iodine seed implantation, ablation, bronchial arterial chemoembolization (BACE) therapy], or received immunotherapy during the first-line standard treatment.
* The patient is accompanied by other malignant tumors and had not been cured.
* White blood cell < 3×10*9/L, absolute value of neutrophils < 1.5×10*9/L, neutrophil/lymphocyte ratio ≥ 3, platelet count < 50×10*9/L, hemoglobin concentration < 90 g/L.
* Liver and kidney dysfunction (creatinine > 176.8 μmol/L; aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 times the upper limit of normal).
* Uncorrectable coagulopathy or active hemoptysis.
* Patient with active infections requires antibiotic treatment.
* Patient has uncontrollable hypertension, diabetes, and cardiovascular disease with obvious symptoms.
* Allergy to contrast agents.
* Women with pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | The time from enrollment to tumor progression or death from any cause, whichever came first, measured in "months", assessed up to 2 years.
  The most common primary endpoint in cancer trials.

SECONDARY OUTCOMES:
Overall Survival | Time from randomization to death from any cause, in "months", assessed up to 2 years. For patients who are still alive at the time of data analysis, OS is calculated based on the date when the patient is last known to be alive.
  The best efficacy endpoint in cancer clinical trials.
Time to tumor untreatable progression | The time interval between randomization to tumor progression that patients are unable to further receive treatment, assessed up to 12 months.
  End point of antitumor drug trial.
Objective Response Rate | Proportion of patients who achieved complete remission (CR) or partial remission (PR) according to mRECIST criteria, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
Disease Control Rate | Proportion of patients with complete remission (CR), partial remission (PR), and stable disease (SD) according to mRECIST criteria, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
Duration of Overall Response | The time from the first assessment of the tumor as complete remission or partial remission to the first assessment as disease progression or death from any cause, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
Tumor biomarkers | From pre-procedure to every follow-up time, assessed up to 2 years.
  carcinoembryonic antigen, carbohydrate antigen 125, squamous cell carcinoma, etc
Eastern Cooperative Oncology Group Score | From pre-procedure to every follow-up time, assessed up to 2 years.
  The patient's performance status score is divided into 6 grades. The lowest grade is 0, and the highest grade is 5. The patient's physical state deteriorates as the grade rises.
Recurrence rate of hemoptysis | From date of randomization to every follow-up time, assessed up to 2 years.
  Hemoptysis occurs again
Quality of life Questionare-Core score | From date of randomization to every follow-up time, assessed up to 2 years.
  The European Organization for Reasearch and Treatment of Cancer Quality of life Questionare-Core score. All items and subscales were converted from 0 to 100, with higher scores indicating better overall quality of life.
The incidence of adverse events and serious adverse events | From date of randomization to every follow-up time, assessed up to 2 years.
  Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Pain assessment | From date of randomization to every follow-up time, assessed up to 2 years.
  Visual Analogue Scale/Score.The tool is a 10 cm long roving ruler with 11 scales ranging from 0 to 10. A score of 0 means no pain, and a score of 10 means unbearable pain. The higher the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Xihui Ying, MD., Study Director — The Central Hospital of Lishui City

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers.
  Shared data does not provide any private information of the participants.